CLINICAL TRIAL: NCT06524479
Title: Investigating the Functional Characteristics During Wakefulness and Sleep Based on SEEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-208-002
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Refractory Epilepsy; Sleep
Keywords: homeostatic sleep pressure; synaptic plasticity
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — SpeA protein, Streptococcus pyogenes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SEEG recordings and SPES effects (Experimental): Single-pulse electrical stimulation (SPES) evokes transient neuronal responses that propagate through functional networks, providing a powerful tool to map brain connectivity. When delivered at low frequencies (0.05 Hz, every 20 s), SPES allows quantitative assessment of dynamic network interactions while avoiding long-term synaptic modifications. These stimulation-induced responses, recorded via stereoelectroencephalography (SEEG), reveal both local and distributed neural activity with millisecond precision.
  Interventions: Procedure: SEEG recordings and SPES

INTERVENTIONS:
Procedure: SEEG recordings and SPES — This study will utilize stereoelectroencephalography (SEEG) recordings combined with single-pulse electrical stimulation (SPES) to investigate functional brain connectivity and cortical excitability patterns in patients with epilepsy during both wakefulness and sleep states. The SEEG recordings will provide high-resolution intracranial electrophysiological data, while SPES will be employed to actively probe and quantify cortico-cortical connections. This combined approach will enable characterization of state-dependent neural network dynamics.

SUMMARY:
This study aims to collect electrophysiological and clinical data from patients aged 14-65 with drug-resistant epilepsy who underwent SEEG. The collected data will be analyzed to investigate the functional connectivity during wakefulness and sleep states.

DETAILED DESCRIPTION:
Sleep serves as a fundamental physiological state whose disruption has profound implications for neurological health. The daily alternation between sleep and wakefulness reflects an intrinsic circadian rhythm that orchestrates critical fluctuations in cortical excitability and functional connectivity throughout the brain. The cerebral cortex, comprising approximately 80% of total brain volume, forms the neural substrate for higher-order cognitive functions including sensory perception, executive control, and memory processes. Importantly, sleep acts as a global brain modulator that dynamically reorganizes patterns of neural communication across distributed cortical and subcortical networks.

Stereoelectroencephalography (SEEG) provides direct access to intracranial electrophysiological activity with exceptional spatiotemporal resolution. When combined with single-pulse electrical stimulation (SPES), this powerful methodology enables quantitative assessment of inter-regional connectivity through analysis of evoked potentials, allowing precise characterization of both connection strength and directionality. This integrated approach offers unique opportunities to examine how different vigilance states modulate cortical excitability and reorganize functional brain networks, particularly in clinical populations with neurological disorders. The ability to track state-dependent changes in network dynamics provides crucial insights into both normal brain function and pathological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Drug-resistant focal epilepsy
* Justified SEEG exploration in the context of presurgical assessment of epilepsy
* Subjects will be a part of the epilepsy-monitoring unit for long-term SEEG recordings and analysis
* Written non-opposition to study participation

Exclusion Criteria:

* Pregnant women (Contraindication to SEEG exploration)
* Subjects that experience surgical complications during the implant procedure will be excluded from the study

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2026-06-07 (Estimated); Study Completion 2027-10-08 (Estimated)

PRIMARY OUTCOMES:
SEEG recordings with SPES during daytime and sleeptime | 48 hours
  Single-pulse electrical stimulation (SPES) serves as an effective dynamic marker for mapping functional brain connectivity. The stimulation parameters were set at 0.05 Hz, single biphasic pulses, 90 μs per phase, 4 mA.

SECONDARY OUTCOMES:
Dynamic melatonin levels | 48 hours
  Collection of melatonin during the day (12 times a day: at 9:00 am, 10:00 am, 11:00 am, 2:00pm, 3:00pm, 4:00pm, 5:00pm, 7:00pm, 8:00pm, 9:00pm, 10:00pm , 11:00pm and 12:00pm) with salivette measurement. Salivary melatonin was measured by radioimmunoassay.
Dynamic cortisone levels | 48 hours
  Collection of salivary cortisone during the day (12 times a day: at 9:00 am, 10:00 am, 11:00 am, 2:00pm, 3:00pm, 4:00pm, 5:00pm, 7:00pm, 8:00pm, 9:00pm, 10:00pm , 11:00pm and 12:00pm) with salivette measurement.
Dynamic 11-Deoxycortisol levels | 48 hours
  Collection of salivary 11-Deoxycortisol during the day (12 times a day: at 9:00 am, 10:00 am, 11:00 am, 2:00pm, 3:00pm, 4:00pm, 5:00pm, 7:00pm, 8:00pm, 9:00pm, 10:00pm , 11:00pm and 12:00pm) with salivette measurement.
Dynamic 21-Deoxycortisol levels | 48 hours
  Collection of salivary 21-Deoxycortisol during the day (12 times a day: at 9:00 am, 10:00 am, 11:00 am, 2:00pm, 3:00pm, 4:00pm, 5:00pm, 7:00pm, 8:00pm, 9:00pm, 10:00pm , 11:00pm and 12:00pm) with salivette measurement.
Dynamic 18-Hydroxycortisol levels | 48 hours
  Collection of salivary 18-Hydroxycortisol during the day (12 times a day: at 9:00 am, 10:00 am, 11:00 am, 2:00pm, 3:00pm, 4:00pm, 5:00pm, 7:00pm, 8:00pm, 9:00pm, 10:00pm , 11:00pm and 12:00pm) with salivette measurement.
Dynamic 18-Oxocortisol levels | 48 hours
  Collection of salivary 18-Oxocortisol during the day (12 times a day: at 9:00 am, 10:00 am, 11:00 am, 2:00pm, 3:00pm, 4:00pm, 5:00pm, 7:00pm, 8:00pm, 9:00pm, 10:00pm , 11:00pm and 12:00pm) with salivette measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, Beijing, Beijing Municipality, China